CLINICAL TRIAL: NCT07361666
Title: Impact of Preoperative High-Frequency Ultrasound Cutaneous Lesion Extent Assessment on Excision Margin Positivity in Head and Neck Skin Cancer, and the Relationship Between Preoperative Assessment Methods, Inadequate Excision Margins, and Tumor Recurrence (HFUS-CLEAR)
Brief Title: Impact of Preoperative High-Frequency Ultrasound Cutaneous Lesion Extent Assessment on Excision Margin Positivity in Head and Neck Skin Cancer, and the Relationship Between Preoperative Assessment Methods, Inadequate Excision Margins, and Tumor Recurrence
Acronym: HFUS-CLEAR
Status: Not yet recruiting | Type: Observational
Sponsor: Państwowy Instytut Medyczny Ministerstwa Spraw Wewnętrznych i Administracji (Other Government)
Responsible Party: Sponsor
Other Study IDs: 21/BW/2025
Record Dates: First submitted 2026-01-15; First posted 2026-01-23 (Actual); Last update posted 2026-01-23 (Actual); Status verified 2026-01

CONDITIONS: Basal Cell Carcinoma of Skin; Cutaneous Squamous Cell Carcinoma (CSCC); Cutaneous Squamous Cell Carcinoma in Situ (CSCCis); Cutaneous Squamous Cell Carcinoma of the Head and Neck; Basal Cell Carcinoma (BCC); Basal Cell Carcinoma of the Head and Neck; Non-Melanoma Skin Cancer (NMSC)
Keywords: Basal Cell Carcinoma; Squamous Cell Carcinoma; Skin Cancer; Skin Neoplasms; Margins of Excision; Positive Surgical Margins; Recurrence; high-frequency ultrasound; HFUS
MeSH Terms: conditions — Carcinoma, Basal Cell; Carcinoma, Squamous Cell; Skin Neoplasms; Margins of Excision; Recurrence | interventions — Dermoscopy

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Biospecimen Retention: Samples Without DNA — Histopathologic samples obtained during standard-of-care surgical treatment will be processed, evaluated, and stored in accordance with routine clinical practice and applicable local regulations. No additional tissue will be collected for the purposes of this study. All specimens will be retained solely within the framework of standard diagnostic procedures and institutional archiving policies, and will not be stored or retained exclusively for research purposes.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- Lesions with tumor extent assessed preoparatively with high-frequency ultrasound and dermoscopy
  Interventions: Diagnostic Test: High-Frequency Ultrasound; Diagnostic Test: Dermoscopy
- Lesions with tumor extent assessed preoparatively with dermoscopy alone
  Interventions: Diagnostic Test: Dermoscopy

INTERVENTIONS:
Diagnostic Test: High-Frequency Ultrasound — High-frequency ultrasound examination of the tumor will be performed using a GE LOGIQ S7 Expert system with an L8-18i-D linear probe (18 MHz). Imaging will include superficial-preset B-mode gray-scale assessment and color Doppler evaluation of lesion vascularity. Standard ultrasound gel will be applied; the probe will be positioned perpendicularly to the skin surface without pressure, avoiding direct contact with the tumor. Images and measurements will be obtained in at least two orthogonal planes. Maximum tumor depth will be recorded as the greatest value measured from the epidermal surface (or granular layer, when visible) to the deepest hypoechoic point of the lesion. When possible, infiltration of deeper structures (e.g., subcutaneous fat, salivary glands, muscle) will also be evaluated.
  Other Names: HFUS; high-frequency ultrasonography
  Groups: Lesions with tumor extent assessed preoparatively with high-frequency ultrasound and dermoscopy
Diagnostic Test: Dermoscopy — All lesions will undergo standard preoperative dermoscopic evaluation performed by a consultant dermatologist, including assessment of tumor extent and marking of dermoscopically visible tumor borders.
  Other Names: Dermatoscopy

SUMMARY:
Non-melanoma skin cancers (NMSC), particularly basal cell carcinoma (BCC) and cutaneous squamous cell carcinoma (cSCC), are the most common malignancies in Caucasians, with the majority of tumors located in the head and neck due to chronic ultraviolet exposure. Although BCC has very low metastatic potential, while cSCC carries a higher risk of nodal spread, both can cause significant local tissue destruction and functional and cosmetic impairment. Complete excision with histologically clear margins remains the standard treatment; however, incomplete or close excision margins are reported in a substantial proportion of cases and are associated with increased risk of local recurrence, need for additional treatment, and higher healthcare costs.

Preoperative dermoscopy improves delineation of lateral tumor borders but does not assess depth of invasion. High-frequency ultrasound (HFUS) is a rapid, non-invasive imaging modality that can visualize superficial skin structures and estimate tumor thickness. Previous studies have suggested good agreement between HFUS and histopathologic depth of invasion, but results are not fully consistent, and HFUS has not yet been incorporated into major guideline recommendations for preoperative assessment of NMSC. Further prospective data are needed to clarify whether HFUS can improve surgical planning and margin control.

This prospective study is designed to assess the impact of adding preoperative HFUS to standard dermoscopic evaluation in head and neck BCC and cSCC. The primary objectives are: (1) to compare the frequency of positive or inadequate (<1 mm) histopathologic excision margins between lesions assessed with dermoscopy alone and those assessed with both dermoscopy and HFUS; and (2) to evaluate 5-year local recurrence rates in relation to preoperative assessment method, histopathologic margin status, and subsequent management of inadequate margins (observation, non-surgical treatment, or scar excision). Secondary and additional objectives include: assessing concordance between HFUS-measured and histopathologic depth of invasion; determining the frequency of residual tumor in scars excised after inadequate margins; evaluating recurrence rate according to the site of inadequate margins (lateral vs deep); and identifying patient-related, tumor-related, surgical, and histopathologic predictors of inadequate margins and recurrence. Approximately 400 lesions (BCC or cSCC of the head and neck) qualified for curative surgical excision will be included. Each lesion will constitute an independent study case. All lesions will undergo preoperative assessment, including clinical evaluation with detailed medical history and dermoscopy; in one cohort, lesions will additionally be evaluated with HFUS. HFUS will be performed with an 18-MHz linear probe, using superficial B-mode and color Doppler. Maximum tumor depth will be recorded from the epidermal surface (or granular layer) to the deepest hypoechoic point, with assessment of potential infiltration of deeper structures when visible. Surgical excision and postoperative care will follow standard clinical practice. Postoperative histopathologic assessment of FFPE tumor samples will record tumor histologic type and subtype, margin status, width, depth of invasion, differentiation, inflammation, elastosis, perineural or vascular invasion, and other routinely assessed diagnostic features. In the event of positive or inadequate excision margins, patients will be referred, after consultation with a dermatologist, for further management (observation, non-surgical treatment, or scar excision), depending on clinical indications and patient preferences. Participation in the study will not influence the primary surgical treatment or any decisions regarding subsequent management.

Patients will be followed for at least 5 years according to current clinical guidelines, with dermoscopic skin examination and documentation of local recurrence and its management. The study aims to determine whether incorporating HFUS into preoperative assessment can reduce the frequency of inadequate histologic margins and improve long-term local control in head and neck NMSC.

ELIGIBILITY:
Inclusion Criteria:

* Cutaneous lesion located in the head and neck region with a preoperative diagnosis of basal cell carcinoma (BCC) or squamous cell carcinoma (SCC), established by dermoscopy or biopsy, and qualified for surgical excision with curative intent.
* patient age of 18 years or older.
* Ability of patient to provide voluntary, informed, written consent for participation in the study.
* Confirmation that the patient has read and understood the Patient Information Sheet.

Exclusion Criteria:

* Excisional biopsies without radical intent.
* Lack of histopathologic confirmation of BCC or SCC in the postoperative specimen (incorrect dermoscopic qualification).
* Inability to perform radical surgical excision due to excessive tumor extent, poor general condition of the patient, or lack of patient consent for surgery.
* Pregnancy.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: This study will include all eligible cutaneous basal cell carcinomas (BCC) and cutaneous squamous cell carcinomas (cSCC) of the head and neck surgically treated at the Department of Otolaryngology. Each eligible lesion will constitute an independent study case. In patients with multiple tumors, each lesion may be included separately if it meets all inclusion criteria. Participation requires informed, written consent from the patient after reviewing the Patient Information Sheet.
Sampling Method: Non-Probability Sample
Enrollment: 400 (Estimated)
Dates: Start 2025-12-23 (Estimated); Primary Completion 2033-11-30 (Estimated); Study Completion 2033-11-30 (Estimated)

PRIMARY OUTCOMES:
Excision Margin Status | Postoperative pathology results (within 30 days after excision)
  Assessment of the frequency of positive or inadequate (defined as positive or <1 mm) histopathologic excision margins in head and neck skin cancer specimens, comparing tumors evaluated preoperatively with dermoscopy alone versus dermoscopy plus high-frequency ultrasound (18 MHz). Margin status will be extracted from postoperative pathology reports.
Five-Year Tumor Recurrence | Up to 5 years after primary tumor excision
  Evaluation of recurrence rates over 5 years based on the preoperative tumor assessment approach (dermoscopy vs. dermoscopy plus HFUS), histopathologic margin status (complete vs. incomplete), and the clinical management chosen in cases of incomplete margins (observation, non-surgical therapies, or scar excision).

SECONDARY OUTCOMES:
Concordance Between HFUS-Measured and Histopathologic Depth of Invasion | Preoperative HFUS assessment and postoperative histopathology (within 30 days)
  Quantitative assessment of concordance coefficient between tumor depth measured preoperatively using high-frequency ultrasound (18 MHz) and depth of invasion reported in postoperative histopathology.
Recurrence Rates According to Site of Incomplete Histopathologic Margins | Up to 5 years after primary tumor excision
  Assessment of whether tumor recurrence rates differ depending on the site of incomplete histopathologic margins recorded in the primary excision - peripheral(lateral) margins vs. deep margin.
Frequency of Residual Tumor Cells in Scar Excision Following Incomplete Margins | Scar excision histopathology (within 90 days after primary excision)
  Determination of the proportion of histopathologic evidence of residual tumor cells in scar tissue removed after incomplete excision margins, based on pathology evaluation of the re-excision specimen.

OTHER OUTCOMES:
Patient-Related and Tumor-Related Risk Factors for Incomplete Margins | Postoperative pathology results (within 30 days after excision)
  Evaluation of potential predictors of incomplete histopathologic margins, including demographic and clinical patient characteristics, comorbidities and medical history (such as immunosuppression, prior organ transplant, prior head and neck radiotherapy, previous skin malignancies and premalignant lesions), tumor growth rate, preoperative clinical tumor features (size, location, poorly defined borders, ulceration, primary vs recurrent lesion), surgical technique and surgical excision margin (assessed macroscopically), and histopathologic features (histologic subtype, depth of invasion, differentiation grade, inflammation, and elastosis). Logistic regression models will be applied.
Patient-Related and Tumor-Related Risk Factors for Tumor Recurrence | Up to 5 years after primary tumor excision
  Evaluation of potential factors associated with 5-year recurrence, including demographic and clinical patient characteristics, comorbidities and medical history (such as immunosuppression, prior organ transplant, prior head and neck radiotherapy, previous skin malignancies and premalignant lesions), tumor growth rate, preoperative clinical tumor features (size, location, poorly defined borders, ulceration, primary vs recurrent lesion), surgical technique and surgical excision margin (assessed macroscopically), and histopathologic features (histologic subtype, depth of invasion, differentiation grade, inflammation, and elastosis). Logistic regression models will be applied.

CONTACTS AND LOCATIONS:
Locations (1):
- National Medical Institute of the Ministry of the Interior and Administration in Warsaw, Warsaw, Masovian Voivodeship, Poland